CLINICAL TRIAL: NCT01792999
Title: Koning Breast CT for Breast Imaging in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Koning (Tianjin) Medical Equipment Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KBCT-CN-001
Record Dates: First submitted 2013-01-16; First posted 2013-02-15 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Breast CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-contrast KBCT (No Intervention): About 187 subjects, who had diagnostic imaging of the breast including mammography and were categorized as Breast Imaging-Reporting and Data System(BIRADS) scores 1, 2, 3, 4, or 5, received KBCT imaging without contrast injection.
- Contrast-enhanced KBCT (Experimental): About 231 subjects, who had diagnostic imaging of the breast including mammography and were scheduled for biopsy or surgery, received contrast-enhanced KBCT imaging of the affected breast before biopsy or surgery.
  Interventions: Device: Contrast-enhanced KBCT

INTERVENTIONS:
Device: Contrast-enhanced KBCT — Contrast-enhanced KBCT includes pre-contrast KBCT scan and post-contrast KBCT scan. After the pre contrast scan is completed, a bolus injection of a low osmolar, nonionic, iodinated 300mg of iodine per mL contrast agent, will be injected at a rate of approximately 2.0 mL/s, for a total injection time of approximately 30-60 seconds. 30-60 seconds after the contrast injection, the post-contrast scan will be acquired.
  Arms: Contrast-enhanced KBCT

SUMMARY:
This study is conducted to compare Koning Breast CT (KBCT) to mammography to evaluate if KBCT can improve the diagnostic accuracy of breast cancer. It will also compare contrast-enhanced KBCT (CE-KBCT) to mammography to evaluate if CE-KBCT can further improve the diagnostic accuracy of breast cancer.

ELIGIBILITY:
Non-contrast KBCT

Inclusion Criteria:

* Females at least 35 years of age of any ethnicity
* Had diagnostic imaging
* Will undergo study imaging no later than two weeks from date of diagnostic mammogram
* Is able to undergo informed consent

Exclusion Criteria:

* Pregnancy
* Lactation
* Subjects with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Subjects who are unable to tolerate study constraints.
* Subjects who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkins disease
* Subjects who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Subjects who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis

Contrast-enhanced KBCT

Inclusion Criteria:

* Females at least 35 years of age of any ethnicity
* Had diagnostic imaging and was determined to have biopsy or surgery
* Will undergo study imaging no later than two weeks from date of diagnostic mammogram
* Is able to undergo informed consent

Exclusion Criteria:

Same as the exclusion criteria as non-contrast KBCT, plus the following:

* Abnormal Glomerular Filtration Rate (GFR)/Blood Urea Nitrogen (BUN) or Creatinine at Pre contrast blood screening
* Previous non-ionic contrast reaction
* History of renal dysfunction/kidney disease
* Diabetes mellitus treated with metformin
* Multiple myeloma
* Dehydration
* History of nephrotoxic medication use
* Hyperthyroidism
* Pheochromocytoma
* Sickle Cell Disease

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2012-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of KBCT, CE-KBCT and Mammography | 1 year
  Efficacy of KBCT, CE-KBCT and Mammography will be assessed based on the sensitivity for detecting breast cancer and the specificity for correctly categorizing non-cancer.

SECONDARY OUTCOMES:
Safety of KBCT, CE-KBCT and Mammography | 1 year
  All enrolled and scanned patients will be included in the safety analysis. Anticipated and unanticipated adverse events will be tabulated according to severity and relation to device.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Ye, MD, PhD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Peihong Wu, MD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality